CLINICAL TRIAL: NCT03642067
Title: Phase A Phase 2 Study Evaluating Response and Biomarkers in Patients With Microsatellite Stable (MSS) Advanced Colorectal Cancer Treated With Nivolumab in Combination With Relatlimab
Brief Title: Study of Nivolumab and Relatlimab in Patients With Microsatellite Stable (MSS) Advanced Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J18119; IRB00173537 (Other: JHM IRB); CA224-068 (Other: other)
Record Dates: First submitted 2018-08-15; First posted 2018-08-22 (Actual); Results first posted 2025-01-28 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Microsatellite Stable (MSS) Colorectal Adenocarcinomas; Colorectal Adenocarcinoma
Keywords: Relatlimab; Nivolumab; Immunotherapy; Anti-PD-1; Anti-LAG-3; Antibody; MSS; PD-L1; Microsatellite stability; Colorectal cancer; Colon cancer; Rectal cancer
MeSH Terms: conditions — Spinocerebellar Degenerations; Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Nivolumab; relatlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A: Composite PD-L1/Mucin (CPM) positive colorectal cancer (Experimental): Participants were pre-screened for CPM score. The CPM score integrates the percent of PD-L1 expression at the tumor interface and the percent of acellular mucin in the tumor area ([%PD-L1 + % acellular mucin]/2) using each participant's primary tumor tissue. A CPM score cutoff of greater than or equal to 15% was used to determine CPM positivity.
  Participants received 480mg Nivolumab and 160mg Relatlimab.
  Interventions: Drug: Nivolumab; Drug: Relatlimab
- Cohort B: Composite PD-L1/Mucin (CPM) negative colorectal cancer (Experimental): Participants were pre-screened for CPM score. The CPM score integrates the percent of PD-L1 expression at the tumor interface and the percent of acellular mucin in the tumor area ([%PD-L1 + % acellular mucin]/2) using each participant's primary tumor tissue. A CPM score cutoff of less than 15% was used to determine CPM negativity.
  Participants received 480mg Nivolumab and 160mg Relatlimab.
  Interventions: Drug: Nivolumab; Drug: Relatlimab
- Cohort C: Colorectal cancer with no biomarker evaluation required (Experimental): Participants were not pre-screened for composite PD-L1/mucin (CPM) score.
  Participants received 480mg Nivolumab and 960mg Relatlimab (dose reduced to 480mg or 160mg).
  Interventions: Drug: Nivolumab; Drug: Relatlimab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab was administered IV on day 1 of each 28 day cycle.
  Other Names: OPDIVO, BMS-936558, anti-PD-1
Drug: Relatlimab — Relatlimab was administered IV on day 1 of each 28 day cycle.
  Other Names: BMS-986016, anti-LAG-3

SUMMARY:
The purpose of this study is to evaluate the safety and clinical activity of nivolumab and relatlimab in patients with metastatic or locally advanced microsatellite stable (MSS) colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* ECOG performance status 0 or 1
* Have metastatic or locally advanced microsatellite stable (MSS) colorectal adenocarcinoma.
* Cohort A: Primary lesion has a composite PD-L1/Mucin (CPM) score ≥ 15%.
* Cohort B: Primary lesion has a composite PD-L1/Mucin (CPM) score < 15%.
* Cohort C: Prior surgical resection of primary tumor. Prospective biomarker evaluation not required.
* Must have received at least one chemotherapy regimen.
* Patients with the presence of at least one measurable lesion using RECIST 1.1.
* Patients must have available archival tissue from the surgical resection of their primary tumor.
* Patient's acceptance of tumor biopsies.
* Life expectancy of greater than 3 months.
* Patients must have adequate organ and marrow function defined by study - specified laboratory tests.
* Documented LVEF ≥ 50% - 6 month prior to drug administration.
* Must use acceptable form of birth control while on study.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Known history or evidence of brain metastases. Patients with previously treated brain metastases may participate if they are stable for 4 weeks prior to beginning treatment, have no new or enlarging brain metastases, and are not using steroids for at least 1 week prior to initiation of study treatment.
* Require any antineoplastic therapy.
* History of prior treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4, or anti-Lag-3 antibodies.
* Had chemotherapy, radiation, or steroids within 14 days prior to study treatment.
* Had any cytotoxic drug within 4 weeks prior to initiation of study treatment.
* Hypersensitivity reaction to any monoclonal antibody.
* Has uncontrolled intercurrent acute or chronic medical illness.
* Has an active known or suspected autoimmune disease.
* Has a diagnosis of immunodeficiency.
* Prior tissue or organ allograft or allogeneic bone marrow transplantation.
* Requires daily supplemental oxygen
* History of interstitial lung disease.
* Requires daily supplemental oxygen.
* Significant heart disease
* History of encephalitis, meningitis, or uncontrolled seizures in the year prior to informed consent.
* Infection with HIV or hepatitis B or C at screening.
* Has an active infection.
* Unable to have blood drawn.
* Patient with uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Woman who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dung Le, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Composite PD-L1/Mucin (CPM) Positive Colorectal Cancer; Cohort B: Composite PD-L1/Mucin (CPM) Negative Colorectal Cancer: Participants received 480mg Nivolumab and 160mg Relatlimab on day 1 of each 28 day cycle.
- Cohort C: Colorectal Cancer With no Biomarker Evaluation Required: Participants received 480mg Nivolumab and 960mg Relatlimab (dose reduced to 480mg or 160mg) on day 1 of each 28 day cycle.
Period: Overall Study
Arm/Group | Cohort A: Composite PD-L1/Mucin (CPM) Positive Colorectal Cancer | Cohort B: Composite PD-L1/Mucin (CPM) Negative Colorectal Cancer | Cohort C: Colorectal Cancer With no Biomarker Evaluation Required
Started (Started = enrolled and received at least one dose of study drug) | 12 | 15 | 32
Completed (Completed = evaluable for the primary endpoint of ORR and underwent at least 1 on study scan) | 12 | 15 | 31
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Composite PD-L1/Mucin (CPM) Positive Colorectal Cancer | Cohort B: Composite PD-L1/Mucin (CPM) Negative Colorectal Cancer | Cohort C: Colorectal Cancer With no Biomarker Evaluation Required | Total
Number analyzed (Participants) | 12 | 15 | 32 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 28 | 51
  >=65 years | 1 | 3 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 17 | 30
  Male | 8 | 6 | 15 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 3
  Not Hispanic or Latino | 11 | 13 | 32 | 56
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 9 | 16
  White | 8 | 9 | 21 | 38
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the number of patients achieving a complete response (CR) or partial response (PR) based on RECIST 1.1 criteria. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions. Participants who discontinue due to toxicity or clinical progression prior to post-baseline tumor assessments will be considered as non-responders. Participants who discontinue for other reasons prior to their first dose of study drug will not included in the analysis.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Composite PD-L1/Mucin (CPM) Positive Colorectal Cancer | Cohort B: Composite PD-L1/Mucin (CPM) Negative Colorectal Cancer | Cohort C: Colorectal Cancer With no Biomarker Evaluation Required
Number analyzed (Participants) | 12 | 15 | 32
Participants | 0 | 1 | 2

2. Secondary Outcome: Number of Participants Experiencing Drug-Related Adverse Events (AEs) Requiring Treatment Discontinuation
Description: Defined using NCI CTCAE v5.0
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Composite PD-L1/Mucin (CPM) Positive Colorectal Cancer | Cohort B: Composite PD-L1/Mucin (CPM) Negative Colorectal Cancer | Cohort C: Colorectal Cancer With no Biomarker Evaluation Required
Number analyzed (Participants) | 12 | 15 | 32
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were evaluated for up to 12 months. All-cause mortality was evaluated for up to 35 months.
Description: This study used the descriptions and grading scales found in the revised National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 for adverse event reporting.
Arm/Group | Cohort A: Composite PD-L1/Mucin (CPM) Positive Colorectal Cancer | Cohort B: Composite PD-L1/Mucin (CPM) Negative Colorectal Cancer | Cohort C: Colorectal Cancer With no Biomarker Evaluation Required
All-Cause Mortality (participants affected / at risk) | 12/12 | 15/15 | 26/32
Serious Adverse Events (participants affected / at risk) | 6/12 | 12/15 | 11/32
Other Adverse Events (participants affected / at risk) | 12/12 | 15/15 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Composite PD-L1/Mucin (CPM) Positive Colorectal Cancer (N=12) | Cohort B: Composite PD-L1/Mucin (CPM) Negative Colorectal Cancer (N=15) | Cohort C: Colorectal Cancer With no Biomarker Evaluation Required (N=32)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 3 (3)
Adrenal Insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Arteriovenous malformation (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 2 (2)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholestatic hepatocellular liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 5 (5) | 4 (4) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Infection, C. Difficile (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection, COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (7)
Obstructive hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pyelonephritis (Renal and urinary disorders) | 1 (3) | 0 (0) | 0 (0)
Rectal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ruptured bowel (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Seizures (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 3 (3) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Composite PD-L1/Mucin (CPM) Positive Colorectal Cancer (N=12) | Cohort B: Composite PD-L1/Mucin (CPM) Negative Colorectal Cancer (N=15) | Cohort C: Colorectal Cancer With no Biomarker Evaluation Required (N=32)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 5 (7) | 9 (12)
Abscess (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Adrenal Insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 3 (3)
Alkaline phosphatase increased (Investigations) | 3 (4) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (6) | 2 (3) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Gastrointestinal disorders) | 2 (2) | 8 (9) | 8 (8)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1)
Ascites (Gastrointestinal disorders) | 3 (4) | 1 (2) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0) | 4 (4)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Belching (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Blood bilirubin increased (Investigations) | 3 (3) | 0 (0) | 2 (2)
Blood in stool (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Blurred vision (Eye disorders) | 2 (2) | 1 (1) | 3 (3)
Cardiac troponin T increased (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Chest Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 7 (7)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 4 (4) | 4 (4) | 7 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (3) | 8 (8)
COVID infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Creatinine increased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 4 (5) | 7 (10)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 3 (4)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Ear blockage (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 3 (3) | 5 (6) | 0 (0)
Edema, Localized (General disorders) | 1 (2) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Fatigue (General disorders) | 4 (4) | 4 (4) | 15 (17)
Fever (General disorders) | 3 (4) | 5 (7) | 4 (4)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 3 (3)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 3 (3)
Hematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Herniated Disk (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 4 (5) | 3 (3) | 2 (3)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 2 (2) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2) | 6 (8)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Infection, H. Pylori (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 4 (4)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (4) | 0 (0) | 0 (0)
Malodorous urine (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Nail changes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 7 (9) | 5 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Nodule, skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 1 (1)
Pain (General disorders) | 3 (4) | 2 (2) | 14 (20)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Pallor (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Papular urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 7 (11)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 5 (6)
Rectal anastomotic leak (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal Bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal tenesmus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Restless Leg Syndrome (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sialorrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 4 (6) | 6 (8) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 2 (3)
Thrush (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1)
Urinary Hesitancy (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 4 (5) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Vision decreased (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 3 (4) | 7 (11)
Weight gain (Investigations) | 2 (2) | 2 (2) | 2 (4)
Weight loss (Investigations) | 5 (5) | 8 (11) | 14 (19)
Thyroid stimulating hormone, increased (Investigations) | 2 (2) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/67/NCT03642067/Prot_SAP_000.pdf